CLINICAL TRIAL: NCT02672254
Title: Investigation "in Vitro" of New Strategies Alternative to Surgery Against Cutaneous Squamous Cell Carcinoma: Topical Chemotherapy Followed by Superficial Radiotherapy.
Brief Title: New Strategies Against Cutaneous Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Silvia Gil Duran, Doctorate, Corporacion Parc Tauli
Other Study IDs: FPT-2016.11
Record Dates: First submitted 2016-01-22; First posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Cutaneous Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A431NS cell cultures from ATCC of human cutaneous squamous carcinoma.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Shams: Samples without any type of treatment
- Samples with 1 treatment: These samples will be treated with only one therapy: chemical agents such as cisplatin or other metallic compounds, or with superficial radiotherapy. These results will help us understand the effectiveness of each treatment by itself on cSCC cells.
- Samples with 2 treatments: These samples will be treated with both, chemical agents followed by superficial radiotherapy. These results will provide us information concerning the effectiveness of both treatments, wich is expected to be enhanced by the concomitant effects.
  Interventions: Radiation: Samples with 2 treatments

INTERVENTIONS:
Radiation: Samples with 2 treatments — Study the concomitant effects between chemo- and radiotherapy by means of cellular techniques.
  Groups: Samples with 2 treatments

SUMMARY:
The gold treatment for local invasive cutaneous squamous cell carcinoma is surgical excision. Nevertheless, surgery is not always an option as a consequence of the age and/or the health status of the patient. One of the objectives of this study is to assess the effects of cisplatin concomitantly with a subsequent low-energy X-rays irradiation in vitro. In order to enhance the effectiveness of this combined treatment, the temporal fractionation of the platinated compound is expected to be performed.

DETAILED DESCRIPTION:
Cutaneous squamous cell carcinoma (cSCC) accounts for the 20% of the most common skin malignancies, i.e. the non-melanoma skin cancer. cSCC is considered one public health problem because of the high costs of its treatment as cSCC are increasing due to a higher sun exposure, as well as more efficient dermatological examinations. In addition, this kind of skin cancer is characterized by a relatively high risk of metastasis.

The gold standard treatment for local invasive cSCC is based on the surgical excision, leading to a 5-years control rate in low-risk patients of 96%. Nevertheless, surgery for local invasive cSCC is not always an option as a consequence of the age and/or the poor health status of the patient. Therefore, ionizing radiation is used as either primary or adjuvant therapy against cSCC in elderly patients or when surgery would be extremely invasive. Although radiotherapy seem to be a promising option, it needs to be improved in order to damage locally the tumor area, thus avoiding damaging secondary effects on healthy tissues. Typical skin radiation sources are based on superficial, orthovoltage X-rays (XR) beams, as well as electron-beam therapy.

In particular, irradiations of local invasive cSCC by using a superficial XR source at kilovoltage (kV) energy permit a local dose deposition within the tumor volume, with a significant smaller penetration capacity with respect to the higher-energy XR sources. Therefore, kV XR sources become a perfect tool for the treatment of superficial lesions, such as the cSCC. The combination of these keV-energy photons with metallic atoms localized in the tumor would enhance the dose deposited locally in the target, improving thus the therapeutic index of the treatment. Among all the chemotherapeutic options available, platinum-based agents, such as cis-diamminedichloroplatinum (II) (cisplatin or cisPt) has become an essential anti-cancer drug with a substantial therapeutic impact against the most carcinomas-like tumors.

The distortion of the structure of the DNA duplex, converts cisPt in a highly toxic agent per se because of its influence on DNA replication, apoptotic death, and inhibition of the major nuclear repair pathway of cisPt-DNA adducts and radiation-induced DNA breaks. However, dose administration is a key limitation due to the high toxicity of this agent. It is for this reason that the lowest cisPt concentration was used in this study, and the expected effectiveness of cisPt on a cSCC cells were enhanced with a subsequent low-energy XR irradiation in an attempt to explore some new therapeutic strategies against local invasive cSCC.

ELIGIBILITY:
Inclusion Criteria:

* human squamous cutaneous carcinoma cell line

Exclusion Criteria:

* contamination

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A431NS human squamous cutaneous carcinoma cell line was obtained from the American Type Culture Collection. A431NS cells were cultured in flasks of 25 cm2 with Dulbecco's Modified Eagle's Medium (DMEM) supplemented with 1% penicillin/streptomycin, and with 10% fetal calf serum to reach confluence. Two hundred thousand cells were seeded per well in 24-well plates, and incubated for 24 hours at 37ºC and 5% CO2.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Study of the effectiveness of each treatment by means of flow cytometry and transmission electron/photon microscopy | 6 months
  The flow cytometry allows us to analyze the proportion of alive, apoptotic and dead (or necrotic) cells after each treatment, whereas miscroscopy techniques would help us detect cell morphology changes either after chemical agents or X-rays.

SECONDARY OUTCOMES:
Study of the effectiveness of both treatments concomitantly by means of flow cytometry and transmission electron/photon microscopy | 6 months
  The flow cytometry allows us to analyze the proportion of alive, apoptotic and dead (or necrotic) cells after both treatments, whereas miscroscopy techniques would help us detect cell morphology changes (even within the cytoplasm and organelles) after the chemical agents and radiation.

IPD SHARING:
Plan to Share IPD: Undecided